CLINICAL TRIAL: NCT04942639
Title: Phase 3, Multi-centre, Prospective, Open, Randomized, in Two Parallel Groups Study to Evaluate Efficacy and Tolerance of Patient's Learning in Self-taking of Prescribed Asthma Maintenance Treatments and Provided by a Robot Named JOE.
Brief Title: Evaluation of Efficacy and Tolerance of JOE on 4 to 11 Years Old Asthmatic Patients of GINA 2,3,4 and 5 Grades
Acronym: JoeCare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ludocare SAS (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Asthma JoeCare; 2021-A00350-41 (Other: ID-RCB)
Record Dates: First submitted 2021-06-17; First posted 2021-06-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Asthma in Children
Keywords: Asthma, Children, Prevention, Severe Asthma Exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Two parallel groups: Standard Asthma Maintenance Treatment (SAMT) vs SAMT + Joe robot (a new DTX)
Who Masked: Outcomes Assessor
Masking Description: Data analysis performed on anonymous database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard + JOE (Experimental): Standard Maintenance Treatment plus JOE robot
  Interventions: Device: JOE
- Standard (No Intervention): Standard maintenance Treatment

INTERVENTIONS:
Device: JOE — Audiovisual support by the robot when taking maintenance treatments at home.
  Arms: Standard + JOE

SUMMARY:
The main objective of this study is to evaluate efficacy and safety of patient's learning in self-taking of prescribed asthma maintenance treatments and provided by JOE (a new DTX), on the number of severe exacerbations in children with an asthma graded 2, 3, 4 and 5 according to GINA classification.

DETAILED DESCRIPTION:
A new device, named JOE, manufactured by Ludocare, is available since 2019 in France. This new device, compact and connected, was designed to be easy to use by children suffering from chronic disease. JOE is a robot designed to improve compliance with asthama maintenance treatments.To confirm efficacy and safety of a patient's learning in self-taking of asthma maintenance treatments provided by JOE, it has been decided to carry out a clinical study in 4 to 11 years old patients and suffering from asthma graded 2, 3, 4 or 5 according to GINA classification. These patients will be recruited by pneumo-pediatricians at hospital or in private practice. The study is a phase 3, multi-center, prospective, open, 2-parallel groups, randomized and controlled study. Each patient will be randomly allocated in one of two studied treatment groups: standard asthma maintenace treatment (group SCT) vs standard asthma maintenance treatment + JOE (a new DTx) (group SCT + JOE). Patients meeting eligible criteria will be included at Day 0 (Visit V0). For each patient the maximal duration of this study will be 12 months. At day 7 a phone call is planned to evaluate patient/parent's motivation and to detect potential technical and/or therapeutic problems. Three visits are planned then after at4 (M4), 8 (M8) and 12 (M12) months.

ELIGIBILITY:
Inclusion Criteria:

* 4-11years old,
* able to use JOE
* persistent uncontrolled asthma, graded 2, 3 , 4 or 5 on GINA classification
* maintenance treatment since at least 3 months
* having given their informed written consent

Exclusion Criteria:

* asthma naïve-treatment child
* without regular follow-up with the investigator
* participating to another interventional study, with another disease, other treatments or planned modification of prescribed treatments that could interfere with studied disease

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the mean number of severe asthma exacerbations per patient between the two treatment groups during the 12-month follow-up. | 12 months
  Evaluation of patient's learning in self-taking of prescribed treatments and provided by robot companion JOE on number of severe exacerbations needing systemic corticoids. Comparison, between both treatment groups, of number of severe exacerbations over 12 months of follow-up.

SECONDARY OUTCOMES:
Effectiveness of the maintenance treatment measured with c-ACT | 12 months
  Effect of the educational support for the patient when taking treatments and provided by the JOE companion robot on the maintenance treatment effectiveness measured with c-ACT score at each visit.
Tolerance to the maintenance treatment evaluated by the number and type of adverse events | 12 months
  Effect of the educational support for the patient when taking treatments and provided by the JOE companion robot on the tolerance of the maintenance treatment evaluated by the number and type of the adverse events declared to the investigator.
Global costs estimation evaluated by price | 12 months
  Evaluation of the global treatment costs, including the treatment of intercurrent events linked to the disease and their possible consequences (unplanned medical consultations, hospitalizations...).

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Cabinet de pneumologie pédiatrique La Fourane, Aix-en-Provence
  - CHU Amiens, Amiens
  - APHP - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHRU Morvan, Brest
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHI Créteil, Créteil
  - Groupe Hospitalier du Havre, Le Havre
  - CH Saint Joseph, Marseille
  - Cabinet Medeo, Montluçon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - APHP - Hôpital Armand Trousseau, Paris
  - APHP - Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No